CLINICAL TRIAL: NCT00208780
Title: Effects of Tetrahydrobiopterin on Blood Pressure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
Keywords: Oxidative Stress; Endothelium
MeSH Terms: conditions — Hypertension | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose-response of oral BH4 (Experimental): Eight subjects received 100 mg of oral BH4 twice a day and 8 received 200 mg twice daily.
  Interventions: Drug: Tetrahydrobiopterin
- Onset & duration of action of oral BH4 (Experimental): Eight hypertensive subjects were assigned to either 5 mg kg-1 day-1 (n=4) or 10 mg kg-1 day-1 (n=4) of BH4, given in two divided doses orally for 8 weeks.
  Interventions: Drug: Tetrahydrobiopterin

INTERVENTIONS:
Drug: Tetrahydrobiopterin
  Arms: Onset & duration of action of oral BH4
Drug: Tetrahydrobiopterin
  Arms: Dose-response of oral BH4

SUMMARY:
Tetrahydrobiopterin (BH4) is a cofactor for the nitric oxide (NO) synthase enzymes, such that its insufficiency results in uncoupling of the enzyme, leading to release of superoxide rather than NO in disease states, including hypertension. We hypothesized that oral BH4 will reduce arterial blood pressure (BP) and improve endothelial function in hypertensive subjects. Oral BH4 was given to subjects with poorly controlled hypertension (BP >135/85 mm Hg) and weekly measurements of BP and endothelial function made. In Study 1, 5 or 10 mg kg-1 day-1 of BH4 (n=8) was administered orally for 8 weeks, and in Study 2, 200 and 400 mg of BH4 (n=16) was given in divided doses for 4 weeks

DETAILED DESCRIPTION:
Problem of Interest:

Blood vessels are lined by a single layer of cells called the endothelium. These cells actively release substances that influence a variety of functions including blood flow in the arteries. Nitric oxide (NO) is among the most important of these substances. Decrease in NO reduces blood vessel size and increases blood pressure (BP). Subjects with hypertension (high blood pressure) and those with a strong family history of hypertension but without high blood pressure also exhibit endothelial dysfunction and decreased NO activity. This abnormality predisposes individuals with high blood pressure to an increased long term risk of adverse cardiovascular events such as heart attack and stroke.

NO is produced in cells by a reaction mediated by the enzyme endothelial nitric oxide synthase (eNOS). Experimental studies performed at Emory University have shown that tetrahydrobiopterin (BH4), a naturally produced substance, is an essential factor for eNOS to be normally active, because in the event of BH4 deficiency, eNOS switches from producing NO to generating oxygen free radicals that increase oxidant stress in blood vessels leading to vascular damage. Moreover, studies have shown that administration of BH4 to animals with hypertension decreases blood pressure.

A recently completed study performed by the researchers at Emory University showed that BH4 pills given twice a day to 8 patients with poorly controlled high blood pressure for eight weeks improved endothelial function and decreased blood pressure without any significant side effects. After stopping BH4, the blood pressure and endothelial function returned to baseline.

Hypertension has also been linked with diastolic heart failure, a condition where the squeeze of the heart is normal but it relaxes abnormally causing shortness of breath, edema and fatigue. Up to one half of cases of heart failure are caused by diastolic heart failure. Recent evidence shows that the lining cells of the heart also produce NO and that this promotes relaxation of the heart. In addition, studies here at Emory have shown that in animals with high blood pressure, NO production in the heart is reduced compared to normals.

How problem will be studied:

The study will consist of three parts:

We, the researchers at Emory University, will recruit patients with hypertension and randomize them to various doses of BH4 to find out what the lowest dose is that produces a significant response This dose will then be used in patients with hypertension who will be randomized to BH4 or a placebo. Patients will be followed for blood pressure response and for markers of endothelial function using ultrasound and for markers of inflammation using blood samples.

Patients from part 2 with evidence of abnormal heart relaxation on echocardiogram will have repeat echocardiograms after drug administration to study the effects of BH4 on heart relaxation.

Advancement in Scientific Knowledge

This study will advance scientific knowledge by looking at the effects of BH4, a naturally occurring substance without known major side effects, on blood pressure. We will also examine the effect of BH4 on NO and relaxation of the heart muscle. Improvement in blood pressure with BH4 will allow this to be an option for treatment of high blood pressure and potentially reducing the complications associated with this condition.

Standard of care:

Currently the standard of care for patients with high blood pressure includes treatment with Food and Drug Administration (FDA) approved medications such as beta-blockers, angiotensin-converting enzyme (ACE) inhibitors, diuretics and calcium-channel blockers to a goal BP of less than 135/85.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients without childbearing potential between the ages of 18 and 75 years
2. History of documented essential hypertension or newly diagnosed hypertension (BP >140 mmHg systolic and/or 90 mmHg diastolic measured on 2 separate occasions)
3. Patients on conventional anti-hypertensive therapy with poorly controlled hypertension (BP >135/85 mmHg). Their anti-hypertensive regimen will remain unchanged throughout the study period. Patients will not need to stop taking their prescribed anti-hypertensives.
4. Controls will be recruited for part 2 of the study. These will be patients who meet the age and childbearing criteria above, who have no history of hypertension, arterial BP of <130 systolic and <85 diastolic, no evidence of diabetes mellitus, total cholesterol <240 and be non-smoking for at least six months.
5. Patients can be at any stage of hypertension. They can be at any performance status. The only requirement will be that they be able to come to scheduled follow up visits either by themselves or with assistance. Patients will need to be able to give informed consent.

Exclusion Criteria:

1. Female subjects with childbearing potential.
2. History of symptomatic coronary or peripheral vascular disease.
3. Known secondary causes for hypertension
4. Severe uncontrolled hypertension (BP >180 mmHg systolic and /or 110 mmHg diastolic).
5. Severe co-morbid conditions which would limit life expectancy to less than 6 months.
6. Patients unable to give informed consent or adhere to the protocol.
7. Patients participating in another study protocol.
8. Patients with organ failure, creatinine >2.5 mg/dL or hepatic enzymes >2X normal
9. Recent (within 6 weeks) alteration of any concomitant therapy.
10. Presence of intercurrent illness
11. Bleeding disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of BH4 on BP

SECONDARY OUTCOMES:
Evaluate the effects of BH4 on vascular function

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Porkert M, Sher S, Reddy U, Cheema F, Niessner C, Kolm P, Jones DP, Hooper C, Taylor WR, Harrison D, Quyyumi AA. Tetrahydrobiopterin: a novel antihypertensive therapy. J Hum Hypertens. 2008 Jun;22(6):401-7. doi: 10.1038/sj.jhh.1002329. Epub 2008 Mar 6. PMID 18322548